CLINICAL TRIAL: NCT05622110
Title: Laparoscopic Incision Closure Following Gynecological Benign Surgeries in Obese Patients
Brief Title: Laparoscopic Incision Closure s in Obese Patients
Acronym: LICOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aya Mohr Sasson, Principle investigator, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-22-0840
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Incision, Surgical
MeSH Terms: conditions — Obesity; Surgical Wound

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The physician doing follow up will be masked to the type of closure in each side
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One abdominal side (Experimental): Arm randomized for adhesive glue closure
  Interventions: Procedure: Adhesive glue closure
- Second abdominal side (Experimental): Arm randomized for subcuticular suture closure
  Interventions: Procedure: Subcuticular closure

INTERVENTIONS:
Procedure: Adhesive glue closure — Incision closure with adhesive glue
  Arms: One abdominal side
Procedure: Subcuticular closure — Incision closure with 3-0 vicryl subcuticular sutures
  Arms: Second abdominal side

SUMMARY:
Several methods for closure of trocar wounds are known in laparoscopic surgery including mostly transcutaneous or subcuticular suture or adhesive paper tape. Studies comparing laparoscopic incision closure in bariatric population are limited .This is a prospective study that will be conducted in a single tertiary medical center. s obese population comprise most of our surgical candidates, and due to the aforementioned, the aim of our study is to compare the outcomes of both techniques in obese women.

DETAILED DESCRIPTION:
Laparoscopic surgery has become the standard of care for surgical procedures across multiple specialties, reducing perioperative complications, accelerating recovery and providing superior cosmetic results. Trocars are used in laparoscopic procedures to provide a portal for the placement of surgical instruments. Typically, three to four or more trocars of different sizes ranging from 5 to 15 mm in diameter are used in abdominal and pelvic surgery.

Several methods for closure of trocar wounds are known in laparoscopic surgery including mostly transcutaneous or subcuticular suture or adhesive paper tape. The skin closure method should aim to keep the skin closely opposed during the hemostatic and inflammatory healing phases until the overlapping proliferative phase is able to provide tensile strength. The choice of technique is often based on the surgeon's personal experience. and is largely dependent on training exposure and local opinion. There is currently no consensus as to the optimal method of closure of the skin following laparoscopic surgery.

Previous meta-analyses examining skin closure methods for all surgical wounds have found suture to have significantly decreased rates of wound dehiscence compared to tissue adhesive. Meta-analysis published recently by Aitchison et al. compared between sutures, tissue adhesives and adhesive paper tape. They reported no difference in patient-evaluated cosmesis, prolonged pain, or patient satisfaction between the three groups. Nevertheless, no data specifically address the obese population.

Port-site trocar incision closure is a challenging procedure in laparoscopic surgeries, particularly in patients with clinically severe (morbid) obesity. Complications related to port-site trocars, even if uncommon, may have severe consequences that can lead to reoperation and permanent damage Studies comparing laparoscopic incision closure in bariatric population are limited. Fecso et al conducted a retrospective cohort study including 1579 bariatric patients, of them 494 were treated with tissue adhesive for skin closure. They reported that the use of tissue adhesive was more common in patients who developed incisional surgical site infection compared with those without incisional surgical site infection (SSI) (54.3 vs. 30.8%, p = 0.003).

Our department usually practice subcuticular and adhesive glue for the closure of laparoscopic incisions, based on surgeon's preference. As obese population comprise most of our surgical candidates, and due to the aforementioned, the aim of our study is to compare the outcomes of both techniques in obese women.

Material and Methods This is a prospective study that will be conducted in a single tertiary medical center. Study population will include all women undergoing gynecologic laparoscopic surgery with BMI of 30 kg/m² or above. Women with connective tissue disease will be excluded from the study.

Intervention:

1. Each woman will undergo both interventions therefore will serve as her own control. All ports up to 8 mm (following robotic or conventional laparoscopy) will be eligible for inclusion in the study. The umbilicus will serve as a reference separating the right and left side incisions. Each side will be closed randomly using one of the two techniques. Randomizing the closure technique will be done based on the serial number given to each woman on recruitment (En block randomization) :

   Odd serial number: Right side - subcuticular suturing, Left side- adhesive glue Even numbers: Right side- adhesive glue, Left side- subcuticular suturing
2. Incisions would be closed by one or the other following techniques: 1- Subcuticular closure- using 4-0 Monocryl suture will be used; 2- Adhesive glue (Dermabond).
3. On follow up visit 2- and 8-weeks post operation - each woman will complete the validated Patient Scar Assessment Questionnaire (PSAQ) on follow-up at 2- and 8-weeks post operation for the right and left side of the abdomen(10). The PSAQ consists of 4 scored subscales: Appearance, Consciousness, Appearance Satisfaction, and Symptom Satisfaction. Each subscale has a set of questions with a 4-point categorical response (1=most favorable, 4=least favorable). The sum of the scores quantifies each subscale.

Demographic and clinical characteristics will be collected from women's medical files. Operative and post-operative data will be collected including: operation duration, estimated blood loss, operation complications (hypotension, bladder gut or vascular perforation), post-operative complications (hemorrhage, endometritis, vascular - thromboembolic event, ileus).

ELIGIBILITY:
Inclusion criteria:

- All women undergoing gynecologic laparoscopic surgery.

Exclusion criteria:

- Connective tissue disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria includes women undergoing bening gynecological surgeries
Enrollment: 53 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Scar Assessment Questionnaire (PSAQ) | From recruitment until 8 weeks post-operation
  The difference in appearance score of the abdominal scars evaluated by the Patient Scar Assessment Questionnaire (PSAQ) between the two techniques reported by the patients at 2 and 8 weeks follow up

SECONDARY OUTCOMES:
Surgical site infection rate | From recruitment until 8 weeks post-operation
  Surgical site infection rate

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr-Sasson, M.D, Principal Investigator — The University of Texas Health Science Center, Houston, TX
Locations (1):
- University of Texas, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andraos Y. Safety and Efficacy of Trocar Port-Site Closure Using a Biological Plug Closure in Laparoscopic Bariatric Surgery: a Prospective Study. Obes Surg. 2022 Nov;32(11):3796-3806. doi: 10.1007/s11695-022-06238-y. Epub 2022 Sep 7. PMID 36071329
- [Background] Pilone V, Di Micco R, Hasani A, Celentano G, Monda A, Vitiello A, Izzo G, Iacobelli L, Forestieri P. Trocar site hernia after bariatric surgery: our experience without fascial closure. Int J Surg. 2014;12 Suppl 1:S83-6. doi: 10.1016/j.ijsu.2014.05.047. Epub 2014 May 23. PMID 24862661
- [Result] Harvey MH, Cahill J, Wastell C. Laparoscopic general surgery. Br J Hosp Med. 1992 May 6-19;47(9):655-62. PMID 1535528
- [Result] Qian LW, Fourcaudot AB, Yamane K, You T, Chan RK, Leung KP. Exacerbated and prolonged inflammation impairs wound healing and increases scarring. Wound Repair Regen. 2016 Jan-Feb;24(1):26-34. doi: 10.1111/wrr.12381. Epub 2016 Jan 12. PMID 26562746
- [Result] Buchweitz O, Wulfing P, Kiesel L. A prospective randomized trial of closing laparoscopic trocar wounds by transcutaneous versus subcuticular suture or adhesive papertape. Surg Endosc. 2005 Jan;19(1):148-51. doi: 10.1007/s00464-004-9043-2. Epub 2004 Nov 18. PMID 15549624
- [Result] Sajid MS, Siddiqui MR, Khan MA, Baig MK. Meta-analysis of skin adhesives versus sutures in closure of laparoscopic port-site wounds. Surg Endosc. 2009 Jun;23(6):1191-7. doi: 10.1007/s00464-009-0373-y. Epub 2009 Mar 5. PMID 19263132
- [Result] Dumville JC, Coulthard P, Worthington HV, Riley P, Patel N, Darcey J, Esposito M, van der Elst M, van Waes OJ. Tissue adhesives for closure of surgical incisions. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD004287. doi: 10.1002/14651858.CD004287.pub4. PMID 25431843
- [Result] Aitchison LP, Chen AZL, Toms C, Sandroussi C, Yeo DA, Steffens D. To stitch or not to stitch: the skin closure of laparoscopic port sites, a meta-analysis. Surg Endosc. 2022 Oct;36(10):7140-7159. doi: 10.1007/s00464-022-09269-9. Epub 2022 May 24. PMID 35610480